CLINICAL TRIAL: NCT07250932
Title: Exploring the Effectiveness of Somatosensory Cognitive Game Intervention on Cognitive and Physical Functions in Older Adults
Brief Title: Exploring the Effectiveness of Somatosensory Cognitive Game Intervention on Cognitive and Physical Functions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: N202509045
Record Dates: First submitted 2025-11-13; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Function

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Somatosensory Cognitive Game Intervention on Cognitive and Physical (Experimental)
  Interventions: Other: somatosensory cognitive game
- Routine care (No Intervention): no Intervention on Cognitive and Physical

INTERVENTIONS:
Other: somatosensory cognitive game — The experimental group will participate in somatosensory cognitive games for 12 weeks, twice a week, about 30 minutes per session.
  Arms: Somatosensory Cognitive Game Intervention on Cognitive and Physical

SUMMARY:
This study investigates the effects of somatosensory cognitive games interventions on older adults' cognitive and physical functions. The investigators plan to recruit up to 100 participants and randomly assign them to a control group or an experimental group. The experimental group will participate in somatosensory cognitive games for 12 weeks, while the control group will receive routine care. Data will be collected via questionnaires to examine whether somatosensory cognitive games can delay declines in cognitive and physical functions in older adults.

DETAILED DESCRIPTION:
This study investigates the effects of somatosensory cognitive games interventions on the cognitive and physical functions of older adults. The investigators plan to recruit 80 participants and randomly assign them to either a control group or an experimental group. The experimental group will participate in somatosensory cognitive games for 12 weeks, twice a week, about 30 minutes per session; the control group will receive usual care without any specific intervention. All participants will complete four questionnaire assessments to examine whether somatosensory cognitive games can slow decline in cognitive and physical functions.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly individuals aged 65 and above.
2. Able to communicate in Chinese (Mandarin or Taiwanese).
3. Voluntarily participate in this study and sign a written consent form.

Exclusion Criteria:

1. Individuals with severe visual impairments or physical mobility disabilities that prevent them from participating in the game activities designed in this study.
2. Individuals diagnosed with severe dementia who are unable to understand or participate in the research process.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | 3 month follow-up
  MoCA is one of the key cognitive function outcomes that investigators expect to improve after somatosensory cognitive games. MoCA assesses six cognitive dimensions, with a total score of 30. A score of 26 or higher is considered normal. MoCA score of ≤24 may indicate a risk of mild cognitive impairment (MCI), while a MoCA score of ≤20 may indicate a risk of dementia.
Color Trails Test (CTT) | 3 month follow-up
  CTT is one of the key cognitive function outcomes that investigators expect to improve after somatosensory cognitive games. CTT is widely used to assess executive function and processing speed. The first part (CTT-1) evaluates visual-motor skills and attention, while the second part of the CTT (CTT-2) assesses sequencing and cognitive flexibility. Scoring is based on the time required to complete the test, with cutoff times of 240 seconds for CTT-1 and 330 seconds for CTT-2. Shorter completion times indicate better executive function and processing speed.

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | 3 month follow-up
  SPPB is another secondary outcome measure that researchers expect to improve after intervention with somatosensory cognitive games. SPPB is mainly used to assess the physical function and mobility of elderly people, with a total score range of 0-12 points, where higher scores indicate better physical function.
Timed Up and Go Test (TUG) | 3 month follow-up
  TUG is another secondary outcome measure that researchers expect to improve after intervention with somatosensory cognitive games. TUG is an assessment tool for evaluating gait and mobility in elderly people. TUG < 10 seconds indicates normal mobility, TUG 11-20 seconds indicates those who can walk independently (but move more slowly), and TUG > 20 seconds indicates those who require assistive devices (such as walkers).